CLINICAL TRIAL: NCT06888531
Title: Prospective Phase II Clinical Study of Neoadjuvant Chemoradiotherapy Combined With PD-1/PD-L1 Inhibitors In the Treatment of Locally Advanced Resectable Esophageal Squamous Cell Carcinoma
Acronym: LA-ESCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA-ESCC-II-01
Record Dates: First submitted 2025-03-05; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Malignant Neoplasm Primary
Keywords: LA-ESCC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Toripalimab: intravenous infusion, 240mg, D1, Q3W, for 2 consecutive doses; or Envorimab: subcutaneous injection, 400mg, D1, Q3W, for 2 consecutive doses. Albumin-bound paclitaxel: intravenous infusion, 50mg/m2, D1, QW, for 5 consecutive doses. Carboplatin: intravenous infusion, AUC=2, D1, QW, for 5 consecutive doses. Radiotherapy: 41.4Gy/1.8Gy/23F, D1-5, 5 times per week.
  Interventions: Combination Product: Neoadjuvant chemoradiotherapy combined with PD-1/PD-L1 inhibitors for the treatment of locally advanced resectable esophageal squamous cell carcinoma

INTERVENTIONS:
Combination Product: Neoadjuvant chemoradiotherapy combined with PD-1/PD-L1 inhibitors for the treatment of locally advanced resectable esophageal squamous cell carcinoma — Toripalimab: intravenous infusion, 240mg, D1, Q3W, for 2 consecutive doses; or Envorimab: subcutaneous injection, 400mg, D1, Q3W, for 2 consecutive doses. Albumin-bound paclitaxel: intravenous infusion, 50mg/m2, D1, QW, for 5 consecutive doses. Carboplatin: intravenous infusion, AUC=2, D1, QW, for 5 consecutive doses. Radiotherapy: 41.4Gy/1.8Gy/23F, D1-5, 5 times per week.
  Other Names: LA-ESCC

SUMMARY:
A prospective trial design was used to evaluate the efficacy and safety of neoadjuvant chemoradiotherapy combined with PD-1/PD-L1 inhibitors in the treatment of locally advanced resectable esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This study is aimed at resectable thoracic esophageal squamous cell carcinoma with clinical stage T1b-2 N+ M0 or T3-4a anyN M0 (AJCC 8th). The primary endpoint of the study is pathological complete response (pCR). A total of 30 patients with locally advanced resectable esophageal squamous cell carcinoma will be enrolled in the trial after providing informed consent and passing the screening process. The treatment regimens include: Toripalimab: intravenous infusion, 240mg, D1, Q3W, for 2 consecutive doses; or Envorimab: subcutaneous injection, 400mg, D1, Q3W, for 2 consecutive doses. Albumin-bound paclitaxel: intravenous infusion, 50mg/m2, D1, QW, for 5 consecutive doses. Carboplatin: intravenous infusion, AUC=2, D1, QW, for 5 consecutive doses. Radiotherapy: 41.4Gy/1.8Gy/23F, D1-5, 5 times per week.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years
2. ECOG performance score 0-1
3. Histologically or pathologically confirmed resectable thoracic esophageal squamous cell carcinoma, clinical stage T1b-2 N+ M0 or T3-4a anyN M0 (AJCC 8th)
4. No prior anti-tumor treatment before surgery
5. At least one measurable lesion (according to RECIST 1.1 criteria).
6. Normal major organ function

Exclusion Criteria:

1. Allergic to the treatment drugs
2. Patients who have received or are currently receiving other chemotherapy, radiotherapy, immunotherapy or targeted therapy
3. Patients with tumors that have invaded major blood vessels as shown by imaging or those judged by the investigator to be highly likely to invade major blood vessels and cause fatal hemorrhage during the subsequent study period
4. Patients with other malignant tumors that require active treatment within 5 years of the study (except for those that have been adequately treated, such as basal cell or squamous cell skin cancer with an expected 5-year survival rate > 90%, cervical carcinoma in situ, and ductal carcinoma in situ of the breast)
5. Patients with active autoimmune diseases or immunodeficiency
6. Patients who are currently using immunosuppressants or systemic hormones for immunosuppression purposes (dose > 10mg/day of prednisone or other equivalent efficacy hormones) and have continued to use them within 2 weeks before enrollment
7. Patients who have received systemic treatment with high-dose antibiotics within the past 2 weeks
8. Patients who have experienced arterial or venous thrombotic events within 6 months before the first administration, including cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral embolism, etc.), deep vein thrombosis and pulmonary embolism
9. Patients with digestive tract diseases or conditions that may affect drug absorption, including but not limited to active gastric and duodenal ulcers, ulcerative colitis or unremoved gastrointestinal tumors with active bleeding, or other conditions judged by the investigator to be likely to cause gastrointestinal bleeding or perforation, and those with multiple factors affecting oral drug administration (such as inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.)
10. Patients with significant cardiovascular diseases, including but not limited to acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; congestive heart failure with New York Heart Association (NYHA) classification ≥ 2; drug-treated ventricular arrhythmias (including QTc interval ≥ 450 ms for men and ≥ 470 ms for women); left ventricular ejection fraction (LVEF) < 50%
11. Patients with active or uncontrolled severe infections (≥ CTCAE5.0 grade 2 infections), including but not limited to hospitalization due to infectious complications, bacteremia or severe pneumonia, and unexplained fever > 38.5°C before the first administration
12. Patients with symptomatic pleural effusion, pericardial effusion or ascites that require frequent drainage as judged by the investigator
13. Patients with liver cirrhosis or active hepatitis; for hepatitis B, HBsAg positive and HBV DNA exceeding the upper limit of normal (1000 copies/ml or 500 IU/ml); patients with a history of hepatitis B virus (HBV) infection or cured HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and the absence of HBsAg, and normal HBV DNA value during the screening period can be included); for hepatitis C, HCV antibody positive and HCV viral load exceeding the upper limit of normal/HCV RNA or HCV Ab test indicating acute or chronic infection. 14. Patients with urine routine test indicating urine protein ≥++, and confirmed 24-hour urine protein quantification > 1.0g

15. Patients with a history of abuse of psychotropic drugs and unable to quit or with mental disorders 16. Patients with pulmonary fibrosis, pneumoconiosis, radiation pneumonitis, drug-induced pneumonia and severe pulmonary function impairment 17. Pregnant women (positive pregnancy test before medication) or women who are breastfeeding 18. Patients who have undergone surgery (excluding biopsy) within 28 days before enrollment in this study or whose surgical incision has not completely healed 19. Patients who have received or plan to receive live attenuated vaccines within 4 weeks before the first dose 20. Patients who have received any other investigational drug treatment or participated in other interventional studies within 4 weeks before signing the informed consent form 21. Patients who, in the judgment of the investigator, are not suitable for inclusion in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | From enrollment to the end of treatment at 2 years
  pCR

SECONDARY OUTCOMES:
Major pathologic response | From enrollment to the end of treatment at 2 years
  MPR

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided